CLINICAL TRIAL: NCT01149018
Title: A Randomized, Double-blind, Placebo-controlled Trial of Oral Tetrahydrocannabinol (∆-9-THC) in Patients With Fibromyalgia
Brief Title: Efficacy Trial of Oral Tetrahydrocannabinol in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Elyad Davidson, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THC-FMS-HMO-CTIL
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Tetrahydrocannabinol; Chronic Widespread Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetrahydrocannabinol (Experimental)
  Interventions: Drug: Tetrahydrocannabinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — Oral solution of THC in concentration of 5mg/0.2ml. Dose regimen: 5mg 2-4 times/day as tolerated.
  Arms: Tetrahydrocannabinol
Drug: Placebo — Orally administered olive oil. Dose: 0.2ml 2-4 times a day as tolerated
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the effectiveness of oral tetrahydrocannabinol in patients suffering from Fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

- Adult (>18y.o) Patient with Fibromyalgia, diagnosed by ACR criteria

Exclusion Criteria:

- Children < 18 years old

Patients with following psychiatric disorders:

* Psychosis or history of acute psychosis
* Schizophrenia
* Bipolar disorder Patients smoking marijuana, using hashish or any other form of cannabis. Patients with history of drug abuse or illicit drug use Patients receiving chronic treatment with strong opioids (Morphine, Oxycodone, Fentanyl, Methadone, Hydromorphone, Buprenorphine, Pethidine). Weak opioids as Tramadol or Propoxyphene will be allowed.

Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Meaningful change in Total score on Fibromyalgia Impact Questionnaire (FIQ) | 8 weeks

SECONDARY OUTCOMES:
Meaningful change in Brief Pain Inventory average pain severity. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Relief Unit, Hadassah Medical Organisation, Jerusalem, Israel